CLINICAL TRIAL: NCT02673424
Title: Comparison of Clinical Outcomes Between Imaging and Physiology-guided Intervention Strategy in Patients With Intermediate Stenosis: Fractional FLow Reserve And IVUS for Clinical OUtcomes in Patients With InteRmediate Stenosis (FLAVOUR)
Brief Title: Fractional FLow Reserve And IVUS for Clinical OUtcomes in Patients With InteRmediate Stenosis
Acronym: FLAVOUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Samsung Medical Center, Sungkyunkwan University School of Medicine (Unknown); Ulsan University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Inje University (Other); KangWon National University Hospital (Other); Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT02673424
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2020-05

CONDITIONS: Stable Angina
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FFR-guided stenting (Active Comparator): Percutaneous coronaryintervention using drug-eluting stent(s) will be performed by FFR-guided strategy.
  Interventions: Procedure: FFR-guided stenting
- IVUS-guided stenting (Active Comparator): Percutaneous coronaryintervention using drug-eluting stent(s) will be performed by IVUS-guided strategy.
  Interventions: Procedure: IVUS-guided stenting

INTERVENTIONS:
Procedure: FFR-guided stenting — The percutaneous coronaryintervention using drug-eluting stent will be indicated according to following criteria in the FFR-guided strategy arm
  * Criteria for revascularization: The FFR ≤ 0.80 will be targeted for PCI
  Arms: FFR-guided stenting
Procedure: IVUS-guided stenting — The percutaneous coronaryintervention using drug-eluting stent will be indicated according to following criteria in the IVUS-guided strategy arm
  * Criteria for revascularization: Minimum lumen area (MLA) ≤ 3mm2 or (MLA ≤ 4mm2 AND Plaque burden >70%)
  Arms: IVUS-guided stenting

SUMMARY:
To compare the safety and efficacy of FFR (fractional flow reserve)-guided percutaneous coronary intervention (PCI) strategy with IVUS (intravascular ultrasound [IVUS])-guided PCI in patients with intermediate coronary stenosis.

DETAILED DESCRIPTION:
1. Study overview This study is a prospective, open-label, randomized, multicenter trial to test the safety and efficacy of physiology- or imaging-guided PCI in patients with intermediate coronary stenosis.

   The primary hypothesis is that FFR-guided strategy will show non-inferior rate of patients-oriented composite outcomes (POCO) at 24 months after randomization, compared with IVUS-guided strategy in patients with intermediate coronary stenosis.
2. Study population and sample size calculation

   Sample Size Calculation Based on the event rates of previous trials, investigators predicted the rates of POCO at 24 months after PCI will be 10% in the FFR-guided arm, and 12% in the IVUS-guided arm.
   * Primary endpoint: patient-oriented composite outcome (a composite of all-cause death, MI, any repeat revascularization) at 24 months after PCI
   * Design: non-inferiority , delta = 2.5%
   * Sampling ratio: FFR-guided strategy : IVUS-guided strategy = 1:1
   * Type I error (α): One-sided 5%
   * Accrual time : 2 years
   * Total time : 4 years (accrual 2 year + follow-up 2 years)
   * Assumption: POCO 10.0% vs. 12.0% in FFR or IVUS-guided strategy, respectively
   * Statistical power (1- β): 90%
   * Primary statistical method : Kaplan-Meier survival analysis with log-rank test
   * Potential withdrawal rates : total 2%
   * Stratification in Randomization: Presence of Diabetes Mellitus (600 patients (35%) will be Diabetic patients, with 300 patients in each group)

   Based on the above assumption, 1,700 patients (850 patients in each group) will be enrolled in this study with consideration of withdrawal rates.
3. Research Materials and Indication for Revascularization For the FFR-guided strategy arm, a pressure-sensor wire system will be used and the criterion for revascularization is FFR ≤ 0.80. Hyperemia will be induced by intravenous infusion of adenosine (140ug/kg/min). For the IVUS-guided strategy arm, the criterion for revascularization is MLA ≤ 3mm2 or [3mm2 < MLA ≤ 4mm2 and plaque burden > 70%].
4. Funding This is an investigator-initiated study with grant support from Boston Scientific. Other than financial sponsorship, the company has no role in protocol development or the implementation, management, data collection, and analysis of this study.
5. Extended Outcome Follow-Up Following the 2-year follow-up period, clinical outcomes will also be collected until September 30, 2024, to assess the long-term outcomes of each treatment group.

ELIGIBILITY:
1. Inclusion Criteria

   * Subject must be ≥ 19 years ② Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic or imaging evaluation and PCI and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

     * Patients suspected with ischemic heart disease ④ Patients with intermediate degree of stenosis (40-70% stenosis by visual estimation) eligible for stent implantation who need FFR or IVUS for further evaluation ⑤ Target vessel size > 2.5mm

       * Target lesions located at the proximal to mid part of coronary artery
2. Exclusion Criteria

   * Known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Adenosine.

     * Active pathologic bleeding

       * Gastrointestinal or genitourinary major bleeding within the prior 3 months.

         * History of bleeding diathesis, known coagulopathy (including heparin-induced thrombocytopenia) ⑤ Non-cardiac co-morbid conditions with life expectancy < 2 years ⑥ Target lesion located in coronary arterial bypass graft ⑦ Target lesion located in the left main coronary artery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Actual)
Dates: Start 2016-06; Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient-oriented composite outcome | 24 months
  a composite of all death, myocardial infarction (MI) or any revascularization
Long-term patient-oriented composite outcome | Up to 7 years
  A composite of all death, myocardial infarction [MI, including peri-procedural MI] or any revascularization during the extended follow-up period after randomization according to the ARC consensus.

SECONDARY OUTCOMES:
Patient-oriented composite outcome | 12 months
  a composite of all death, myocardial infarction (MI) or any
Stent-oriented composite endpoint | 12 months
  a composite of cardiac death, target-vessel MI, or target lesion revascularization
Stent-oriented composite endpoint | 24 months
  a composite of cardiac death, target-vessel MI, or target lesion revascularization
Cost-effectiveness analysis | 24 months
  medical expenses of treatment and follow-up. Cost estimates utilize micro-costing, the total cost by identifying the utilization of medical resources used, and macro-costing, medical expenses resulting from clinical events from health insurance data.
All-cause death | 24 months
  death from any cause
Cardiac death | 24 months
  death from cardiaccause
Target-vessel and all-cause nonfatal myocardial infarction without per-procedural myocardial infarction | 24 months
  Myocardial infarction during 24 months follow-up without periprocedural myocardial infarction
Target-vessel and all-cause nonfatal myocardial infarction with per-procedural myocardial infarction | 24 months
  Myocardial infarction during 24 months follow-up with periprocedural myocardial infarction
Peri-procedural MI using referred definitions | At discharge (1 week after index procedure)
  Number of participants with peri-procedural myocardial infarction after PCI
Target vessel/lesion revascularization | 24 months
  Number of participants and vessels/lesions with ischemia-driven or any reavascularizations at target vessel/lesion
Non-target vessel/lesion revascularization | 24 months
  Number of participants and vessels/lesions with ischemia-driven or any reavascularizations at non-target vessel/lesion.
Any revascularization | 24 months
  Number of participants and vessels/lesions with ischemia-driven or any revascularizations at any vessel/lesion
Academic Research Consortium defined - Stent thrombosis | 24 months
  Number of participants with definite/probable/possible stent thrombosis
Stroke | 24 months
  Number of participants with ischemic or hemorrhagic stroke
Acute success of procedure | immediately after the intervention
  Device-related, lesion-related and procedure-related success of index procedure (residual diameter stenosis<50% and thrombolysis in myocardial infarction flow 3)
Angina severity measured with Seattle Angina Questionnaires | 12 months
  Seattle Angina Questionnaires (physical limitation and angina frequency were classified as minimal: 75-100, mild: 50-74, moderate: 25-49, severe: 0-24)
Angina severity measured with Seattle Angina Questionnaires | 24 months
  Seattle Angina Questionnaires (physical limitation and angina frequency were classified as minimal: 75-100, mild: 50-74, moderate: 25-49, severe: 0-24)
Long-term patient-oriented composite outcome in subgroups by use of anti-platelet agent and lipid-lowering agents | Up to 7 years
  A composite of all death, myocardial infarction [MI, including peri-procedural MI] or any revascularization during the extended follow-up period in subgroups stratified by use of anti-platelet agent and lipid-lowering agents
Long-term patient-oriented composite outcome in subgroups by lipid profiles | Up to 7 years
  Long-term patient-oriented composite outcome in subgroups stratified by changes in LDL-cholesterol, HDL-cholesterol, and triglyceride during the extended follow-up period
Long-term mortality | Up to 7 years
  All-cause and cardiac death during the extended follow-up period
Long-term myocardial infarction | Up to 7 years
  Myocardial infarction during the extended follow-up period
Long-term any revascularization | Up to 7 years
  Any revascularization during the extended follow-up period
Long-term target vessel failure | Up to 7 years
  Target vessel failure (cardiac death, target vessel MI, target vessel revascularization) during the extended follow-up period
Long-term target vessel myocardial infarction | Up to 7 years
  Target vessel myocardial infarction during the extended follow-up period
Long-term target vessel revascularization | Up to 7 years
  Target vessel revascularization during the extended follow-up period
Long-term target lesion revascularization | Up to 7 years
  Target lesion revascularization during the extended follow-up period
Long-term non-target lesion revascularization-target vessel revascularization | Up to 7 years
  Non-target lesion revascularization-target vessel revascularization during the extended follow-up period
Long-term stent thrombosis | Up to 7 years
  Stent thrombosis (definite/probable/possible) during the extended follow-up period
Long-term stroke | Up to 7 years
  Stroke (ischemic and hemorrhagic) during the extended follow-up period
Landmark analysis for patient-oriented composite outcome | Up to 7 years
  A 2 year landmark analysis of patient-oriented composite outcome and its individual outcome components
Long-term patient-oriented composite outcome in the medical treatment group | Up to 7 years
  Patient-oriented composite outcome and individual components of outcomes in the medical treatment group
Long-term patient-oriented composite outcome in the PCI group | Up to 7 years
  Patient-oriented composite outcome and individual components of outcomes in the PCI group
Long-term patient-oriented composite outcome according to PCI optimization | Up to 7 years
  Patient-oriented composite outcome and individual outcome components among patients in the PCI group, comparing those who received PCI optimization to those who did not.
Landmark analysis for target vessel failure | Up to 7 years
  A 2 year landmark analysis of target vessel failure and its individual outcome components
Long-term target vessel failure in the medical treatment group | Up to 7 years
  Target vessel failure and individual components of outcomes in the medical treatment group
Long-term target vessel failure in the PCI group | Up to 7 years
  Target vessel failure and individual components of outcomes in the PCI group
Long-term target vessel failure according to PCI optimization | Up to 7 years
  Target vessel failure and individual outcome components among patients in the PCI group, comparing those who received PCI optimization to those who did not.
Long-term target vessel failure according to IVUS-derived plaque characteristics | Up to 7 years
  Target vessel failure (cardiac death, target vessel MI, target vessel revascularization) during the extended follow-up period according to IVUS-derived plaque characteristics
Long-term target vessel failure according to QFR values | Up to 7 years
  Target vessel failure (cardiac death, target vessel MI, target vessel revascularization) during the extended follow-up period according to QFR values

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital; Seung-Jea Tahk, MD, PhD, Principal Investigator — Ajou University School of Medicine; JianAn Wang, MD, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (5):
- The Second Affiliated Hospital, School of Medicine, Zhejiang University, Zhejiang, China
- South Korea (4):
  - Keimyung University Dongsan Medical Center, Daegu
  - Inje University Ilsan Paik Hospital, Goyang
  - Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Seoul National University Hospital, Seoul, Korea, Seoul

IPD SHARING:
Plan to Share IPD: Yes
The deidentified data will be shared after publication of first manuscript
Supporting Information: Study Protocol
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Derived] Ding D, Zhang J, Wu P, Wang Z, Shi H, Yu W, Hu X, Kang J, Hahn JY, Nam CW, Doh JH, Lee BK, Kim W, Huang J, Jiang F, Zhou H, Chen P, Tang L, Jiang W, Chen X, He W, Ahn SG, Yoon MH, Kim U, Ki YJ, Shin ES, Tahk SJ, Pu J, Wijns W, Wang J, Koo BK, Tu S. Prognostic Value of Postpercutaneous Coronary Intervention Murray-Law-Based Quantitative Flow Ratio: Post Hoc Analysis From FLAVOUR Trial. JACC Asia. 2025 Jan 7;5(1):59-70. doi: 10.1016/j.jacasi.2024.10.019. eCollection 2025 Jan. PMID 39886193
- [Derived] Hwang D, Kim HL, Ko J, Choi H, Jeong H, Jang SA, Hu X, Kang J, Zhang J, Jiang J, Hahn JY, Nam CW, Doh JH, Lee BK, Kim W, Huang J, Jiang F, Zhou H, Chen P, Tang L, Jiang W, Chen X, He W, Ahn SG, Kim U, Ki YJ, Shin ES, Kim HS, Tahk SJ, Wang J, Lee TJ, Koo BK; FLAVOUR Investigators. Cost-effectiveness of Fractional Flow Reserve Versus Intravascular Ultrasound to Guide Percutaneous Coronary Intervention: Results From the FLAVOUR Study. Korean Circ J. 2025 Jan;55(1):34-46. doi: 10.4070/kcj.2024.0156. Epub 2024 Oct 11. PMID 39601394
- [Derived] Lee JH, Ahn SG, Jeon HS, Lee JW, Youn YJ, Zhang J, Hu X, Wang J, Lee JM, Hahn JY, Nam CW, Doh JH, Lee BK, Kim W, Huang J, Jiang F, Zhou H, Chen P, Tang L, Jiang W, Chen X, He W, Yoon MH, Tahk SJ, Kim U, Ki YJ, Shin ES, Hwang D, Kang J, Kim HS, Koo BK. Discordance Between Angiographic Assessment and Fractional Flow Reserve or Intravascular Ultrasound in Intermediate Coronary Lesions: A Post-hoc Analysis of the FLAVOUR Trial. Korean Circ J. 2024 Aug;54(8):485-496. doi: 10.4070/kcj.2024.0046. Epub 2024 Jun 10. PMID 38956940
- [Derived] Lee JM, Kim H, Hong D, Hwang D, Zhang J, Hu X, Jiang J, Nam CW, Doh JH, Lee BK, Kim W, Huang J, Jiang F, Zhou H, Chen P, Tang L, Jiang W, Chen X, He W, Kang J, Ahn SG, Yoon MH, Kim U, Ki YJ, Shin ES, Choi KH, Park TK, Yang JH, Song YB, Choi SH, Gwon HC, Koo BK, Kim HS, Tahk SJ, Wang J, Hahn JY; FLAVOUR Investigators. Clinical Outcomes of Deferred Lesions by IVUS Versus FFR-Guided Treatment Decision. Circ Cardiovasc Interv. 2023 Dec;16(12):e013308. doi: 10.1161/CIRCINTERVENTIONS.123.013308. Epub 2023 Nov 29. PMID 38018840
- [Derived] Koo BK, Hu X, Kang J, Zhang J, Jiang J, Hahn JY, Nam CW, Doh JH, Lee BK, Kim W, Huang J, Jiang F, Zhou H, Chen P, Tang L, Jiang W, Chen X, He W, Ahn SG, Yoon MH, Kim U, Lee JM, Hwang D, Ki YJ, Shin ES, Kim HS, Tahk SJ, Wang J; FLAVOUR Investigators. Fractional Flow Reserve or Intravascular Ultrasonography to Guide PCI. N Engl J Med. 2022 Sep 1;387(9):779-789. doi: 10.1056/NEJMoa2201546. PMID 36053504